CLINICAL TRIAL: NCT02267824
Title: The Effects of Extraoral Photobiomodulation on the Rate of Orthodontic Alignment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biolux Research Holdings, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OP2
Record Dates: First submitted 2014-10-10; First posted 2014-10-20 (Estimated); Results first posted 2016-03-15 (Estimated); Last update posted 2018-08-27 (Actual); Status verified 2018-08

CONDITIONS: Malocclusion
Keywords: Alignment phase; Photobiomodulation; Orthodontic treatment; Malocclusion; OrthoPulse™
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Extraoral OrthoPulse® PBM (Experimental): Subjects assigned to this group receive full mouth fixed orthodontic appliance treatment in conjunction with receiving daily extraoral OrthoPulse® photobiomudulation (PBM) treatments.
  Interventions: Device: Extraoral OrthoPulse® PBM; Other: Fixed Orthodontic Appliance Treatment
- Orthodontic Treatment (Control) (Other): Subjects assigned to this group receive full mouth fixed orthodontic appliance treatment, only.
  Interventions: Other: Fixed Orthodontic Appliance Treatment

INTERVENTIONS:
Device: Extraoral OrthoPulse® PBM — Patients carry out daily extraoral OrthoPulse® PBM treatments at home.
  Arms: Extraoral OrthoPulse® PBM
Other: Fixed Orthodontic Appliance Treatment — Patients are treated for full mouth fixed orthodontic appliance treatment by the qualified Principal Investigator (PI). Orthodontic treatment procedures carried out per the traditional practices of the PI and dental office.

SUMMARY:
The aim of this study is to determine if extraoral OrthoPulse®, which emits extraoral LED (Light Emitting Diode) photobiomodulation (PBM), reduces the time it takes to complete orthodontic alignment.

ELIGIBILITY:
Inclusion Criteria:

* Permanent dentition
* Class I malocclusion with irregularity score of greater than 2 mm in either arch
* Good oral hygiene

Exclusion Criteria:

* Any medical or dental condition that could potentially affect study results
* Patients currently using any investigational drug or any other investigational device
* Patients planning to relocate or move during the treatment period
* Use of bisphosphonates
* Pregnant females

Ages: 11 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 101 (Actual)
Dates: Start 2010-12; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chung H Kau, DDS, Principal Investigator — University of Alabama (UAB) Birmingham
Locations (4):
- United States (2):
  - Department of Orthodontics, School of Dentistry, University of Alabama, Birmingham, Alabama
  - Shaughnessy Orthodontics, Suwanee, Georgia
- Clinique Dentaire Alvaro de la Fuente, L'Ile Perrot, Quebec, Canada
- Department of Orthodontics, Faculty of Dentistry, Mahidol University, Bangkok, Thailand

REFERENCES:
- [Background] Nimeri G, Kau CH, Corona R, Shelly J. The effect of photobiomodulation on root resorption during orthodontic treatment. Clin Cosmet Investig Dent. 2014 Jan 15;6:1-8. doi: 10.2147/CCIDE.S49489. eCollection 2014. PMID 24470774
- [Background] Ekizer A, Uysal T, Guray E, Akkus D. Effect of LED-mediated-photobiomodulation therapy on orthodontic tooth movement and root resorption in rats. Lasers Med Sci. 2015 Feb;30(2):779-85. doi: 10.1007/s10103-013-1405-3. Epub 2013 Aug 29. PMID 23990217
- [Background] Ekizer A, Uysal T, Guray E, Yuksel Y. Light-emitting diode photobiomodulation: effect on bone formation in orthopedically expanded suture in rats--early bone changes. Lasers Med Sci. 2013 Sep;28(5):1263-70. doi: 10.1007/s10103-012-1214-0. Epub 2012 Nov 9. PMID 23139069
- [Background] Uysal T, Ekizer A, Akcay H, Etoz O, Guray E. Resonance frequency analysis of orthodontic miniscrews subjected to light-emitting diode photobiomodulation therapy. Eur J Orthod. 2012 Feb;34(1):44-51. doi: 10.1093/ejo/cjq166. Epub 2010 Dec 27. PMID 21187526
- [Background] El-Bialy T, Alhadlaq A, Felemban N, Yeung J, Ebrahim A, Hassan AH. The effect of light-emitting diode and laser on mandibular growth in rats. Angle Orthod. 2015 Mar;85(2):233-8. doi: 10.2319/030914-170.1. Epub 2014 Jul 14. PMID 25017014
- [Background] Kau CH, Kantarci A, Shaughnessy T, Vachiramon A, Santiwong P, de la Fuente A, Skrenes D, Ma D, Brawn P. Photobiomodulation accelerates orthodontic alignment in the early phase of treatment. Prog Orthod. 2013 Sep 19;14:30. doi: 10.1186/2196-1042-14-30. PMID 24326198
- [Background] Dias FJ, Issa JP, Vicentini FT, Fonseca MJ, Leao JC, Siessere S, Regalo SC, Iyomasa MM. Effects of low-level laser therapy on the oxidative metabolism and matrix proteins in the rat masseter muscle. Photomed Laser Surg. 2011 Oct;29(10):677-84. doi: 10.1089/pho.2010.2879. Epub 2011 Jul 11. PMID 21745137
- [Background] Silveira PC, Silva LA, Fraga DB, Freitas TP, Streck EL, Pinho R. Evaluation of mitochondrial respiratory chain activity in muscle healing by low-level laser therapy. J Photochem Photobiol B. 2009 May 4;95(2):89-92. doi: 10.1016/j.jphotobiol.2009.01.004. Epub 2009 Jan 21. PMID 19232497
- [Background] Cruz DR, Kohara EK, Ribeiro MS, Wetter NU. Effects of low-intensity laser therapy on the orthodontic movement velocity of human teeth: a preliminary study. Lasers Surg Med. 2004;35(2):117-20. doi: 10.1002/lsm.20076. PMID 15334614
- [Background] Esper MA, Nicolau RA, Arisawa EA. The effect of two phototherapy protocols on pain control in orthodontic procedure--a preliminary clinical study. Lasers Med Sci. 2011 Sep;26(5):657-63. doi: 10.1007/s10103-011-0938-6. Epub 2011 May 31. PMID 21626017
- [Background] Youssef M, Ashkar S, Hamade E, Gutknecht N, Lampert F, Mir M. The effect of low-level laser therapy during orthodontic movement: a preliminary study. Lasers Med Sci. 2008 Jan;23(1):27-33. doi: 10.1007/s10103-007-0449-7. Epub 2007 Mar 15. PMID 17361391
- [Background] Sousa MV, Scanavini MA, Sannomiya EK, Velasco LG, Angelieri F. Influence of low-level laser on the speed of orthodontic movement. Photomed Laser Surg. 2011 Mar;29(3):191-6. doi: 10.1089/pho.2009.2652. Epub 2011 Jan 23. PMID 21254890
- [Background] Heravi F, Moradi A, Ahrari F. The effect of low level laser therapy on the rate of tooth movement and pain perception during canine retraction. Oral Health Dent Manag. 2014 Jun;13(2):183-8. PMID 24984620
- [Background] Whelan HT, Smits RL Jr, Buchman EV, Whelan NT, Turner SG, Margolis DA, Cevenini V, Stinson H, Ignatius R, Martin T, Cwiklinski J, Philippi AF, Graf WR, Hodgson B, Gould L, Kane M, Chen G, Caviness J. Effect of NASA light-emitting diode irradiation on wound healing. J Clin Laser Med Surg. 2001 Dec;19(6):305-14. doi: 10.1089/104454701753342758. PMID 11776448
- [Background] Weber JB, Pinheiro AL, de Oliveira MG, Oliveira FA, Ramalho LM. Laser therapy improves healing of bone defects submitted to autologous bone graft. Photomed Laser Surg. 2006 Feb;24(1):38-44. doi: 10.1089/pho.2006.24.38. PMID 16503787
- [Background] Saito S, Shimizu N. Stimulatory effects of low-power laser irradiation on bone regeneration in midpalatal suture during expansion in the rat. Am J Orthod Dentofacial Orthop. 1997 May;111(5):525-32. doi: 10.1016/s0889-5406(97)70152-5. PMID 9155812
- [Background] Masha RT, Houreld NN, Abrahamse H. Low-intensity laser irradiation at 660 nm stimulates transcription of genes involved in the electron transport chain. Photomed Laser Surg. 2013 Feb;31(2):47-53. doi: 10.1089/pho.2012.3369. Epub 2012 Dec 16. PMID 23240874
- [Background] Oron U, Ilic S, De Taboada L, Streeter J. Ga-As (808 nm) laser irradiation enhances ATP production in human neuronal cells in culture. Photomed Laser Surg. 2007 Jun;25(3):180-2. doi: 10.1089/pho.2007.2064. PMID 17603858
- [Background] Sun X, Zhu X, Xu C, Ye N, Zhu H. [Effects of low energy laser on tooth movement and remodeling of alveolar bone in rabbits]. Hua Xi Kou Qiang Yi Xue Za Zhi. 2001 Oct;19(5):290-3. Chinese. PMID 12539482

RESULTS

PARTICIPANT FLOW:
Groups:
- Extraoral OrthoPulse® PBM: Subjects assigned to this group receive full mouth fixed orthodontic appliance treatment in conjunction with receiving daily extraoral OrthoPulse® PBM treatments.
- Orthodontic Treatment (Control): Subjects assigned to this group receive full mouth fixed orthodontic appliance treatment only.
Period: Overall Study
Arm/Group | Extraoral OrthoPulse® PBM | Orthodontic Treatment (Control)
Started | 83 | 18
Completed | 73 | 17
Not Completed | 10 | 1
Not completed — Pregnancy | 1 | 1
Not completed — Lost to Follow-up | 4 | 0
Not completed — Protocol Violation | 3 | 0
Not completed — Did Not Meet Initial Dental Criteria | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Extra-Oral OrthoPulse™: Subjects assigned to this group receive full mouth fixed orthodontic appliance treatment by the qualified Principal Investigator (PI), in conjunction with receiving daily extra-oral OrthoPulse™ treatments. Treatment and follow-up appointments per the traditional practices of the PI and dental office.
  Extra-Oral OrthoPulse™: Patients carry out daily extra-oral OrthoPulse™ treatments at home.
- Control: Subjects assigned to this group receive only full mouth fixed orthodontic appliance treatment by the qualified Principal Investigator (PI), and no extra-oral OrthoPulse™ treatments. Treatment and follow-up appointments per the traditional practices of the PI and dental office.
- Total: Total of all reporting groups
Arm/Group | Extra-Oral OrthoPulse™ | Control | Total
Number analyzed (Participants) | 83 | 18 | 101
Age, Customized [Mean (Standard Deviation); unit: years]
  Age | 18.0 (7.0) | 19.5 (7.4) | 18.3 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 12 | 68
  Male | 27 | 6 | 33
Region of Enrollment [Number; unit: participants]
  Canada | 13 | 0 | 13
  United States | 49 | 9 | 58
  Thailand | 21 | 9 | 30

OUTCOME MEASURES:

1. Primary Outcome: Rate of Orthodontic Anterior Alignment in Millimetres Per Week (mm/wk) by Means of Little's Irregularity Index (LII) for Extraoral OrthoPulse® PBM and Non-OrthoPulse® PBM Treated Patients.
Time Frame: Participants followed for the time it takes to complete orthodontic anterior alignment, an expected average of 30-120 days from the start of orthodontic treatment, depending on the severity of the case.
Measure: Mean (Standard Deviation); unit: millimeters per week (mm/wk)
Groups:
- Extraoral OrthoPulse® PBM and Orthodontic Treatment: Subjects assigned to this group receive full mouth fixed orthodontic appliance treatment in conjunction with receiving daily extraoral OrthoPulse® PBM treatments.
Arm/Group | Extraoral OrthoPulse® PBM and Orthodontic Treatment | Orthodontic Treatment (Control)
Number analyzed (Participants) | 73 | 17
millimeters per week (mm/wk) | 1.12 (1.05) | 0.49 (0.40)

ADVERSE EVENTS:
Arm/Group | Extraoral OrthoPulse® PBM | Orthodontic Treatment (Control)
Serious Adverse Events (participants affected / at risk) | 0/83 | 0/18
Other Adverse Events (participants affected / at risk) | 1/83 | 0/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Extraoral OrthoPulse® PBM (N=83) | Orthodontic Treatment (Control) (N=18)
Cheek redness (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No